CLINICAL TRIAL: NCT03372473
Title: Safety and Efficacy of Montelukast + Loratadine vs. Montelukast for the Control of Mild to Moderate Persistent Asthma in Children: Randomized Controlled Clinical Trial
Brief Title: Montelukast and Loratadine in Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: National Institute of Pediatrics, Mexico (Other Government); Laboratorios Senosiain, S.A. de C.V. (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Translational Research Center on Mother-Child Health, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Montelukast2017
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Loratadine; montelukast

STUDY DESIGN:
Intervention Model Description: Randomized clinical crossover trial, in 80 children who were allocated to receive montelukast + loratadine vs montelukast in two different periods of 4 weeks each, with a 2 weeks of wash-out between periods of treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Children allocated on different arms will receive montelukast + loratadine vs. montelukast + placebo. Both product are identical in appearence and flavor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast mixed with Loratadine (Experimental): Montelukast 5mg mixed with Loratadine 5mg one dose a day
  Interventions: Drug: Montelukast mixed with Loratadine
- Montelukast (Active Comparator): Montelukast 5mg one dose per day
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast mixed with Loratadine — Montelukast 5mg mixed with Loratadine 5mg, one dose per day
  Arms: Montelukast mixed with Loratadine
Drug: Montelukast — Montelukast 5mg
  Arms: Montelukast

SUMMARY:
Randomized controlled trial in 80 children with mild to persistent moderate asthma, who were randomized to receive montelukast 5mg + loratadine 5mg vs. montelukast 5mg + placebo for loratadine to evaluate the efficacy in terms of improvement of symptoms. Secondary outcome was the days off without the use of rescue medication; reduction of levels of cysteinyl leukotrienes (Cys-LTS), nitric oxide (FeNO), intracellular adhesion molecule type 1 (ICAM-1) and interleukin 8 (IL-8) in condensed exhaled air; the improvement of day and night symptoms; the reduction in the frequency of night awakenings; the improvement in the quality of life; the percentage of related adverse events; the need to use systemic steroids; the number of visits to the emergency department secondary to the presence of an asthma attack; the number of hospitalizations secondary to asthma attacks; and the improvement in the percentage of FEV1 in relation to the predicted.

DETAILED DESCRIPTION:
Asthma is a disease with increasing prevalence worldwide that produces significant deterioration of the quality of life in children and development of important complications and economic, social impact. Considering the concept of a common airway (coexistence of asthma and rhinitis), joint management initiatives with anti-asthmatics and anti-histamines have been published. The primary objective of this clinical trial is to evaluate the efficacy and safety of the use of montelukast + loratadine in children with asthma on the improvement of symptoms and secondarily to evaluate the impact on a) the days off without the use of rescue medication; b) reduction of levels of cysteinyl leukotrienes (Cys-LTS), nitric oxide (FeNO), intracellular adhesion molecule type 1 (ICAM-1) and interleukin 8 (IL-8) in condensed exhaled air; c) the improvement of day and night symptoms; d) the reduction in the frequency of night awakenings; e) the improvement in the quality of life; f) the percentage of related adverse events; g) the need to use systemic steroids; h) the number of visits to the emergency department secondary to the presence of an asthma attack; i) the number of hospitalizations secondary to asthma attacks; and j) the improvement in the percentage of FEV1 in relation to the predicted. We included 80 children from 6 to 12 years old, any sex, with mild to moderate persistent asthma, after signing an informed consent letter by parents or guardians or signing the child's consent (> 8 years). Children with chronic diseases associated with the disease of interest were excluded (heart disease, nephropathy, liver disease of any kind); with any other lung disease other than asthma; with a history of hypersensitivity to montelukast or loratadine or with a history of concomitant use of medications that interact significantly with montelukast or loratadine

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 12 years old
* Any sex
* Persistent mild to moderate asthma
* Signature of informed consent letter by parents or guardians
* Letter of assent of the minor for children over 9 years of age

Exclusion Criteria:

* Chronic pathologies associated with the disease of interest (heart disease, nephropathy, liver disease of any kind)
* Any other lung disease other than asthma
* History of hypersensitivity to montelukast or loratadine
* Concomitant use of medications that interact significantly with montelukast or loratadine

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Free of symptoms | 10 weeks
  Number of days free of symptoms associated to asthma episodes

SECONDARY OUTCOMES:
Free of rescue medication | 10 weeks
  Number of days free for use of rescue medications
Reduction of airway inflammatory profile | 10 weeks
  Measurement of inflamatory biomarkers in exhaled respiratory air
Reduction of awakenings | 10 weeks
  Frequency of nocturn awakenings
Quality of Life | 10 weeks
  Changes in PedsQL during the treatment
Emergency visits | 10 weeks
  Number of emergency visits secondary to asthma crisis
Adverse Events | 10 weeks
  Frequency of reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez Castrellon, MD, Principal Investigator — Hospital General Dr. Manuel Gea Gonzalez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Result] Carpagnano GE, Spanevello A, Sabato R, Depalo A, Palladino GP, Bergantino L, Foschino Barbaro MP. Systemic and airway inflammation in sleep apnea and obesity: the role of ICAM-1 and IL-8. Transl Res. 2010 Jan;155(1):35-43. doi: 10.1016/j.trsl.2009.09.004. PMID 20004360
- [Result] Carraro S, Corradi M, Zanconato S, Alinovi R, Pasquale MF, Zacchello F, Baraldi E. Exhaled breath condensate cysteinyl leukotrienes are increased in children with exercise-induced bronchoconstriction. J Allergy Clin Immunol. 2005 Apr;115(4):764-70. doi: 10.1016/j.jaci.2004.10.043. PMID 15805996
- [Result] Zanconato S, Carraro S, Corradi M, Alinovi R, Pasquale MF, Piacentini G, Zacchello F, Baraldi E. Leukotrienes and 8-isoprostane in exhaled breath condensate of children with stable and unstable asthma. J Allergy Clin Immunol. 2004 Feb;113(2):257-63. doi: 10.1016/j.jaci.2003.10.046. PMID 14767439
- [Result] Massingham K, Fox S, Smaldone A. Asthma therapy in pediatric patients: a systematic review of treatment with montelukast versus inhaled corticosteroids. J Pediatr Health Care. 2014 Jan-Feb;28(1):51-62. doi: 10.1016/j.pedhc.2012.11.005. Epub 2013 Jan 9. PMID 23312367
- [Result] Corren J, Manning BE, Thompson SF, Hennessy S, Strom BL. Rhinitis therapy and the prevention of hospital care for asthma: a case-control study. J Allergy Clin Immunol. 2004 Mar;113(3):415-9. doi: 10.1016/j.jaci.2003.11.034. PMID 15007339